CLINICAL TRIAL: NCT00552370
Title: A Randomized, Open-Label, Parallel-Design Trial. Glycemia Optimization Treatment: Safety of Glucose Control Using Dosing Algorithms With Lantus®(Insulin Glargine [rDNA Origin[) in Adult Individuals With Type 2 Diabetes.
Brief Title: Glycemic Optimization Treatment Study
Acronym: GOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4045
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Lantus®

SUMMARY:
To compare the frequency of severe hypoglycemia events for 5 dosing algorithms of Lantus®, each of varying intensity and defined by their end-of -study target for self monitored plasma glucose(SMPG), in patients with Type 2 diabetes mellitus, with inadequate glycemic control (A1C greater than or equal to 7.0%) on oral antidiabetic drug therapy(OAD).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give their signed informed consent.
2. Diagnosis of Type 2 DM for at least 6 months.
3. Males and females greater than or equal to 18 years of age.
4. A1c greater than or equal to 7.0%.
5. Current (last 2 months) diabetes therapy with oral anti-hyperglycemia agents only.
6. Demonstrated willingness and ability to inject insulin glargine.
7. Able to understand and willing to comply with procedures required by the protocol and have access to a phone.
8. Demonstrated ability and willingness to perform self-monitoring of blood glucose (SMBG) and use of the algorithm calculator (AL-CAL).
9. BMI greater than 25.0 kg/m2.
10. Subjects who, in the opinion of the investigator, should be initiated on insulin therapy.

Exclusion Criteria:

1. Cardiac status New York Heart Association (NYHA) III-IV (Appendix A).
2. For subjects treated with metformin (Glucophager, Glucophage XRr, Glucovancer, Metaglipr , or Avandametr) plus a serum creatinine greater than 1.5 mg/dL (133 μmol/L) for males or greater than 1.4 mg/dL (124 μmoL) for females, the inability or unwillingness to discontinue these medications, and to remain off them through the entire study.
3. For subjects on thiazolidinediones, the inability or unwillingness to discontinue these medications and to remain off them through the entire study.
4. Planned pregnancy, pregnancy, or lactation.
5. Serum creatinine greater than 3.0 mg/dL (266 μmol/L).
6. Serum glutamic pyruvic transaminase (SGPT) greater than 2.5 x the upper limit of normal range.
7. Any current malignancy or cancer within the past 5 years (except adequately treated basal cell carcinoma or cervical carcinoma in situ).
8. Diagnosis of dementia or mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
9. Hypersensitivity to Lantus® insulin or any of its components.
10. Any disease or condition, including the abuse of illicit drugs, prescription medicines, or alcohol that, in opinion of the sponsor/investigator, may interfere with the completion of the study.
11. Current (last 2 months) insulin therapy.
12. With the exception of thiazolidinediones (for all potential subjects) and for subjects who are taking metformin and have an exclusionary creatinine level, the ability or unwillingness to continue pre-study anti-hyperglycemia agents at pre-study dosages through the entire study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5062 (Actual)
Dates: Start 2003-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To compare the frequency of severe hypoglycemia events for 5 dosing algorithms of Lantus®, each of varying intensity and defined by their end-of-study target for self monitored blood glucose (SMBG). | From the start to the end of the study

SECONDARY OUTCOMES:
To compare the number of subjects whose final A1c is <7.0% at the end of the study for the 5 dosing algorithms. | From the start to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, Study Director — Sanofi